CLINICAL TRIAL: NCT00405977
Title: The Effect of Magnesium Sulphate on the Time Course of Rocuronium Induced Neuromuscular Block - A Randomised Electrophysiology Study
Brief Title: The Effect of Magnesium Sulphate on the Time Course of Rocuronium Induced Neuromuscular Block
Acronym: MagRoc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Christoph Czarnetzki, Study Leader, University Hospital, Geneva
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER 05-055
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Neuromuscular Blockade
Keywords: Neuromuscular block; Magnesium; Rocuronium; Time course of action
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiologic saline (Placebo Comparator)
  Interventions: Drug: Physiologic saline
- Magnesium sulphate (Active Comparator)
  Interventions: Drug: Magnesium sulphate

INTERVENTIONS:
Drug: Physiologic saline — Intravenous infusion of the study solution, 1 ml per kg bodyweight, corresponding to MgSO4 60 mg kg-1 in the magnesium group and 1 ml per kg physiological saline. The infusion will be given with during 15 minutes.
  Arms: Physiologic saline
Drug: Magnesium sulphate — Intravenous infusion of the study solution, 1 ml per kg bodyweight, corresponding to MgSO4 60 mg kg-1 in the magnesium group. The infusion will be given during 15 minutes.
  Arms: Magnesium sulphate

SUMMARY:
The aim of this study is to investigate whether an optimized pre-treatment with intravenous magnesium enhances the speed of onset of a standard intubation dose of rocuronium.

DETAILED DESCRIPTION:
In a previous study pre-treatment with intravenous MgSO4 60 mg kg-1 was not shown to have any impact on the onset of action of rocuronium [Kussmann et al, 1997]. Yet, in that study, MgSO4 was injected as a bolus after induction of anaesthesia, one minute only before the injection of the neuromuscular blocking agent. We suppose that magnesium needs some time to penetrate the neuromuscular endplate and to shift the Mg/Ca ratio in favor of magnesium. Thus, the particular design of the previous study may explain why magnesium had no scope to enhance the speed of onset of action of rocuronium.

The aim of our study is to investigate whether an optimised pre-treatment with magnesium (short infusion rather than bolus injection; reasonable delay between administration of magnesium and subsequent injection of the neuromuscular blocking agent) enhances the speed of onset of a standard intubation dose of rocuronium.

1. Preanaesthetic preparation

   * Solid food and liquid intake will not be allowed for a minimum of six hours before induction
   * Patients will be premedicated with 7.5 mg oral midazolam 45 min prior to induction
   * Standard monitoring will consist of: ECG, SaO2, ETCO2, non-invasive blood pressure, rectal or oesophageal T°
2. Study drug administration

   * Intravenous infusion of the study solution, 1 ml per kg bodyweight, corresponding to MgSO4 60 mg kg-1 in the magnesium group. The infusion will be given with an Infusomat during 15 minutes.
3. Induction and maintenance of anaesthesia

   * At the end of the study drug infusion, and after a preoxygenation period of three minutes, anaesthesia will be induced with sufentanil 0.2µg kg-1 and propofol, using a Target Controlled Infusion (TCI) system (Base Primea, Fresenius-Vial, Brezins, France) and the pharmacokinetic model of Schnider et al [Schnider et al, 1999]. The initial effect site concentration will be 4 µg ml-1.
   * Maintenance of anaesthesia will be with a propofol effect site
4. Neuromuscular monitoring

   * Neuromuscular function will be monitored using the TOF Watch® SX (NV Organon) and TOF nerve stimulation. The guidelines for good clinical research practice in pharmacodynamic studies of NMBAs will be followed.
   * The ulnar nerve is stimulated through surface electrodes, and the adductor pollicis muscle response is measured.
   * After the stabilisation period, rocuronium 0.6 mg kg-1 (2 x ED95) will be injected intravenously during 5 seconds.
   * The trachea will be intubated after a 95% depression of the first twitch

5.1. Neuromuscular measurements

* Onset time = time from beginning of injection of rocuronium until a 95% depression of the first twitch (T1).
* Duration 25% = time from beginning of injection of rocuronium until 25% T1 recovery.
* Recovery index T25-75 = time between 25% T1 recovery and 75% T1 recovery.
* Clinical recovery T25 - 0.9 = time between 25% T1 recovery and TOF ratio (T1/T4) of 0.9 (corresponding to safe extubation condition).

5.2. Haemodynamics

* Blood pressure
* Heart rate These measurements will be done before (baseline), and at 5-minute intervals during the study drug infusion. Before and immediately after tracheal intubation, haemodynamic measurements will be repeated.

5.3. Adverse events, safety

* Any minor adverse event (no need for intervention) or major adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiology (ASA) status I or II
* Adults, aged 18 years to 60 years
* Scheduled for elective surgery lasting longer than 120 min without need for continuous curarisation

Exclusion Criteria:

* A history of allergy or hypersensitivity to rocuronium
* Neuromuscular disease
* Preoperative medications known to influence neuromuscular function (for instance, certain antibiotics and anticonvulsants)
* Electrolyte abnormalities
* Hepatic or renal insufficiency
* Patients with a body mass index <19 or >28 kg m2
* Pregnant or breastfeeding women
* Expected difficult intubation or mask ventilation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To study whether a pre-treatment with MgSO4, 60 mg kg-1, administered as an intravenous infusion 15 minutes prior to induction enhances the speed of onset of a standard intubation dose of rocuronium | 1 to 5 minutes
  Onset time ist the time in seconds from start of injection of rocuronium until 95% depression of the first twitch (T1) of the Train of four (TOF)

SECONDARY OUTCOMES:
To study whether, and to what extent, pre-treatment with MgSO4 prolongs recovery characteristics of the neuromuscular block that is induced by rocuronium | minutes to hours
To study possible haemodynamic effects of pre-treatment with MgSO4. | hours

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Czarnetzki, MD, MBA, Principal Investigator — University Hospital of Geneva, Anesthesia Department; Martin Tramer, MD, PhD, Study Chair — University Hospital of Geneva, Anesthesia Department
Locations (1):
- University Hospital of Geneva, Anesthesia Department, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Result] Czarnetzki C, Lysakowski C, Elia N, Tramer MR. Time course of rocuronium-induced neuromuscular block after pre-treatment with magnesium sulphate: a randomised study. Acta Anaesthesiol Scand. 2010 Mar;54(3):299-306. doi: 10.1111/j.1399-6576.2009.02160.x. Epub 2009 Nov 16. PMID 19919585